CLINICAL TRIAL: NCT05498935
Title: Prolonged Cardiopulmonary Bypass (CPB) Time as a Predictive Factor for Acute Gastrointestinal Injury (AGI) After Heart Valve Replacement
Brief Title: Prolonged Cardiopulmonary Bypass Time as a Predictive Factor for AGI After Heart Valve Replacement
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, Professor of Surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: CPB-AGI
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Heart Valve Diseases
Keywords: Heart valve diseases; Gastrointestinal tract
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CPB time ≥ 90 minutes: No intervention, regular therapy
  Interventions: Other: CPB time
- CPB time < 90 minutes: No intervention, regular therapy
  Interventions: Other: CPB time

INTERVENTIONS:
Other: CPB time — Cardiopulmonary bypass time

SUMMARY:
In this retrospective study, the investigators will analyze the correlation between cardiopulmonary bypass (CPB) time and acute gastrointestinal injury (AGI), and the outcomes of AGI in patients undergoing heart valve replacement.

DETAILED DESCRIPTION:
Patients with heart valve diseases often have chronic cardiac insufficiency. Patients undergoing heart valve replacement with CPB are always complicated with gastrointestinal tract ischemia-reperfusion injury, which usually leads to AGI. AGI after cardiovascular surgery, especially in that use CPB, is associated with significant morbidity and an increase in peri-operative mortality. Prolonged CPB time could be predictive of AGI following heart valve replacement. This study is to analyze the correlation between CPB time and AGI, and the outcomes of AGI in patients undergoing heart valve replacement. The investigators hope that the benefits will include fewer patients becoming seriously postoperative AGI and mortality after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing heart valve replacement surgery with CPB
* Age > 18 years and ≤ 70 years

Exclusion Criteria:

* Patients combined with severe hematological disease, respiratory disease, and other critical diseases
* Patients had severe disorder of multiple systems and organs or severe pulmonary hypertension
* Have received major gastrointestinal surgery within 5 years
* Inflammatory bowel disease (IBD), including ulcerative colitis, Crohn's disease, or colitis
* Acute gastroenteritis
* Clostridium difficile or Helicobacter pylori infection
* Chronic constipation
* Peptic ulcer
* Polyps in the stomach or intestines
* Gastrointestinal neoplasms
* Abdominal hernia
* Irritable bowel syndrome
* Acute or chronic cholecystitis, hepatitis
* Patients who died during surgery
* Patients with digestive system tumors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart valve diseases
Sampling Method: Non-Probability Sample
Enrollment: 1070 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary bypass (CPB) time | 1 month
  Was defined it as the sum of times of CPB during surgery (minutes).
The AGI score | 1 month
  The AGI score of the patient within the seventh postoperative day was performed according to the European Society of critical care (2012) guidelines for AGI.

SECONDARY OUTCOMES:
Number of bowel sounds | 1 month
  The return time of bowel sounds was evaluated morning and evening.
First defecation time | 1 month
  The time to the first defecation was asked morning and evening after surgery
Proportion of cocci and bacilli in feces | 1 month
  The first feces were collected in sterile containers for the bacterial smear
Alanine aminotransferase (ALT) | 1 month
  We defined it as the maximum value of ALT within 7 days after surgery.
Aspartate aminotransferase (AST) | 1 month
  We defined it as the maximum value of AST within 7 days after surgery
Left ventricular ejection fraction (LVEF) | 1 month
  We measured the LVEF on the 1st and 3rd days after operation by echocardiographic examinations

CONTACTS AND LOCATIONS:
Overall Officials: Wenbo Meng, M.D. Ph.D, Principal Investigator — LanZhou University
Locations (1):
- Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: Undecided
If patients permitted

REFERENCES:
- [Result] Gallitto E, Sobocinski J, Mascoli C, Pini R, Fenelli C, Faggioli G, Haulon S, Gargiulo M. Fenestrated and Branched Thoraco-abdominal Endografting after Previous Open Abdominal Aortic Repair. Eur J Vasc Endovasc Surg. 2020 Dec;60(6):843-852. doi: 10.1016/j.ejvs.2020.07.071. Epub 2020 Aug 24. PMID 32855033
- [Result] Buchbinder A, Adler H, Ballard H. An unusual and unreported toxicity to erythropoietin. Am J Hematol. 1993 Apr;42(4):412-3. doi: 10.1002/ajh.2830420428. No abstract available. PMID 8494005